CLINICAL TRIAL: NCT02722863
Title: Post Marketing Surveillance Study of Safety and Efficacy of Samsca® Tablets Under the "New Drug Re-Examination"
Brief Title: Samsca Post Marketing Surveillance Study
Acronym: Samsca PMS
Status: Completed | Type: Observational
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 156-KOA-1201n
Record Dates: First submitted 2016-03-18; First posted 2016-03-30 (Estimated); Results first posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-02

CONDITIONS: Hypervolemic and Euvolemic Hyponatremia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This Post-Marketing Surveillance will be conducted in accordance with the local regulation of New Drug Re-examination. The surveillance will be conducted for 6 years of the re-examination period (01Sep2011~31Aug2017). Each subject will be observed at least for 4 days during the surveillance period.

DETAILED DESCRIPTION:
This study will be conducted as a prospective, single-arm, multicenter study. Findings on examination, diagnosis, opinions and observations implemented as per general medical practice during the observational period will be documented in the case report forms by the investigators or responsible staffs at the institution since the surveillance is an observational study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study :

  1. Patients who have hyponatremia in euvolemic or hypervolemic states, defined as serum sodium level < 125 mEq/L or hyponatremia that is symptomatic and has resisted correction with fluid restriction
  2. Patients who are prescribed Samsca® treatment as per investigator's medical judgment
  3. Patients who gave written authorization to use their personal and health data
  4. Patients starting Samsca® treatment after agreement is in place Investigators will refer to the product market authorization (label) for inclusion criteria.

Exclusion Criteria:

* Subjects presenting with any of the following will not be included in the study:

  1. Patients who have been treated with Samsca®
  2. Patients with known or suspected hypersensitivity to tolvaptan or to any ingredient of the drug
  3. Patients requiring urgent intervention to raise serum sodium acutely.
  4. Inability of the patient to sense or appropriately respond to thirst.
  5. Hypovolemic hyponatremia
  6. Concomitant use of strong CYP3A inhibitors
  7. Anuric patients
  8. Volume depletion patients
  9. Hypernatremia patients
  10. Women who are pregnant or possibly pregnant and lactation
  11. Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption Investigators will refer to the product market authorization (label) for exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The treatment of clinically significant hypervolemic and euvolemic hyponatremia [serum sodium < 125 mEq/L or hyponatremia that is symptomatic and has resisted correction with fluid restriction], including patients with heart failure, cirrhosis, Syndrome of Inappropriate Antidiuretic Hormone (SIADH) and etc.
Sampling Method: Probability Sample
Enrollment: 908 (Actual)
Dates: Start 2013-07-09 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - Bong Seng Hospital, Busan
  - Daegu Catholic University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chung-Ang University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Samsca: Patients who have hyponatremia in euvolemic or hypervolemic states, defined as serum sodium level < 125 mEq/L or hyponatremia that is symptomatic and has resisted correction with fluid restriction.
  Patients who are prescribed Samsca® treatment as per investigator's medical judgment Patients who gave written authorization to use their personal and health data Patients starting Samsca® treatment after agreement is in place
Period: Overall Study
Arm/Group | Samsca
Started | 908
Completed | 908
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: all patients who received Samsca® tablets at least once and had at least one post-treatment assessment during the study in approved indication and dosage regimen
Groups:
- Safety Set: all patients who received Samsca® tablets at least once and had at least one post-treatment assessment during the study in approved indication and dosage regimen
Arm/Group | Safety Set
Number analyzed (Participants) | 668
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 154
  >=65 years | 514
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 326
  Male | 342
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Safety Measure
Description: Adverse Events (AEs)
Time Frame: 4days
Population: Safety analysis set was defined as all patients who received Samsca® tablets at least once and had at least one post-treatment assessment during the study in approved indication and dosage regimen.
Measure: Number (95% Confidence Interval); unit: percentage of AE
Groups:
- Safety Set: a safety evaluation was conducted on 668 patients out of 908 patients' collected survey
Arm/Group | Safety Set
Number analyzed (Participants) | 668
percentage of AE | 17.37 [14.57 to 20.46]

2. Secondary Outcome: Change of the Serum Sodium Level(mEq/L) at the First Visit and Day 4 After the First Visit
Description: In the efficacy analysis set, mean change of serum sodium level (mEq/L)on the 4th day compared to the first visit
Time Frame: Follow-up at least 4 days after first Samsca® dose
Population: the efficacy set is patients who received Samsca® tablets for at least 4 consecutive days and had the data on serum sodium level(mEq/L) on the 4th day of receiving Samsca® tablets.
Measure: Mean (Standard Deviation); unit: mean change of serum sodium level(mEq/L)
Groups:
- Efficacy Set: patients who received Samsca® tablets for at least 4 consecutive days and had the data on serum sodium level(mEq/L) on the 4th day of receiving Samsca® tablets.
Arm/Group | Efficacy Set
Number analyzed (Participants) | 452
mean change of serum sodium level(mEq/L)
  Firtst visit | 123.78 (4.81)
  4th day | 134.83 (5.69)

ADVERSE EVENTS:
Time Frame: up to 4 days.
Arm/Group | Safety Set
All-Cause Mortality (participants affected / at risk) | 6/668
Serious Adverse Events (participants affected / at risk) | 10/668
Other Adverse Events (participants affected / at risk) | 110/668
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Set (N=668)
Azotaemia (Renal and urinary disorders) | 2 (2)
Pyelonephritis (Renal and urinary disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Condition aggravated (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac failure (Vascular disorders) | 1 (1)
Bilirubinaemia (Hepatobiliary disorders) | 1 (1)
Heart valve disorders (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Set (N=668)
Constipation (Gastrointestinal disorders) | 43 (55)
Diarrhoea (Gastrointestinal disorders) | 16 (16)
Nausea (Gastrointestinal disorders) | 10 (11)
Vomiting (Gastrointestinal disorders) | 8 (8)
Abdominal pain (Gastrointestinal disorders) | 6 (6)
Indigestion (Gastrointestinal disorders) | 4 (5)
Mouth dry (Gastrointestinal disorders) | 4 (5)
Mucosal ulceration (Gastrointestinal disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Tongue discolouration (Gastrointestinal disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (4)
Thirst (Metabolism and nutrition disorders) | 3 (3)
Weight decrease (Metabolism and nutrition disorders) | 3 (3)
Hypernatraemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Polydipsia (Metabolism and nutrition disorders) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Weight increase (Metabolism and nutrition disorders) | 1 (1)
Fever (General disorders) | 8 (8)
Back pain (General disorders) | 3 (3)
Pain (General disorders) | 3 (3)
Leg pain (General disorders) | 2 (2)
Oedema peripheral (General disorders) | 2 (2)
Asthenia (General disorders) | 1 (1)
Hyperpyrexia (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Medicine ineffective (General disorders) | 1 (1)
Azotaemia (Renal and urinary disorders) | 5 (5)
Pyelonephritis (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 2 (2)
Cystitis (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Oliguria (Renal and urinary disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4)
Delirium (Psychiatric disorders) | 3 (3)
Anorexia (Psychiatric disorders) | 4 (4)
Anxiety (Psychiatric disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Coughing (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 8 (8)
Hypertension (Vascular disorders) | 4 (4)
Headache (Nervous system disorders) | 6 (6)
Dizziness (Nervous system disorders) | 4 (4)
Hyperkinesia (Nervous system disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1)
Skeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Palpitation (Cardiac disorders) | 2 (2)
Tachycardia ventricular (Cardiac disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1)
ALT increased (Hepatobiliary disorders) | 1 (1)
AST increased (Hepatobiliary disorders) | 1 (1)
Post-operative haemorrhage (Investigations) | 1 (1)
Decubitus ulcer (Investigations) | 1 (1)
Infection (Immune system disorders) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Leucopenia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-20): https://cdn.clinicaltrials.gov/large-docs/63/NCT02722863/Prot_SAP_000.pdf